CLINICAL TRIAL: NCT01624857
Title: Perioperative Statin for Depression in Patients Undergoing Coronary Artery Bypass Surgery
Brief Title: Statin for Depression in Patients Undergoing Coronary Artery Bypass Graft
Acronym: Stress CABG
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 20120618
Record Dates: First submitted 2012-06-17; First posted 2012-06-21 (Estimated); Last update posted 2013-08-15 (Estimated); Status verified 2012-05

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control group (Placebo Comparator): Placebo for at least 5 days before the CABG surgery, then continue to take for a month after the surgery.
  Interventions: Drug: Placebo
- statin group (Active Comparator): Rosuvastatin 20mg/d for at least 5 days before the CABG surgery, then continue to take for a month
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Rosuvastatin — Rosuvastatin for at least 5 days before the CABG surgery, then continue to take for a month after the surgery.
  Arms: statin group
Drug: Placebo — Placebo for at least 5 days before the CABG surgery, then continue to take for a month after the surgery.
  Arms: control group

SUMMARY:
Depression is frequently observed in patients with coronary heart disease (CHD) and represents a significant risk factor for major cardiovascular events. Previous study has proved that high sensitive C-reactive protein (hsCRP) was an independent predictor for depression in CABG patients at 6 months after bypass surgery. Statins can effectively reduce the blood levels of hsCRP. This study aim to examine whether statins can improve the prognosis of depressive patients undergoing coronary artery bypass surgery through reducing the levels of hsCRP.

DETAILED DESCRIPTION:
Depression is frequently observed in patients with coronary heart disease (CHD) and represents a significant risk factor for major cardiovascular events. Depression in patients with existing CHD confers a relative risk between 1.5 and 2.5 for cardiac morbidity and mortality. In previous cross-sectional and prospective studies, the prevalence of major depression in patients with CHD ranged from 10% to 47%, and slightly higher rates were reported (28%) in patients requiring coronary artery bypass grafting (CABG). In CABG patients, symptoms of depression may increase mortality after bypass surgery and were associated with atherosclerotic progression.

In 2008, the American Heart Association recommended routine screening for depression in patients with CHD in various settings, including the hospital, physician's office, clinic, and cardiac rehabilitation center. In recent years, growing evidence also suggests the existence of a bidirectional relationship between depressed mood and inflammation. Dantzer and associates reported that inflammation can lead to the development of symptoms of depression in vulnerable individuals. Consistent with these findings, high-sensitivity C-reactive protein (hsCRP), currently as one available clinical biomarker of inflammation, was reported associated with increased long-term mortality and extended hospital length of stay in patients undergoing nonemergency CABG-only surgery. And our previous study showed that elevated serum hsCRP is an independent predictor for depression in CABG patients not only preoperatively but also up to 6 months after surgery.

This study will enroll patients undergoing coronary artery bypass surgery in Fuwai Hospital. At study entry, participants will be interviewed during their index hospitalization, to collect information about depressive symptoms, functioning, quality of life, and medical care. Demographic characteristics, medical history, clinical features, diagnostic tests, medications, procedures, and in-hospital outcomes of patients will be abstracted from medical records by well trained professional abstractors. At 1 month and 6 month after discharge, participants will return to the clinic for follow up visits, a face-to-face interview will be conducted to get information about clinical events, depressive symptoms, functioning, quality of life, and medical care during the recovery period. Practical guidelines will be established based on the findings to improve patients' outcomes in future finally.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients for coronary artery bypass graft surgery

Exclusion Criteria:

* Previous CABG surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2012-06; Primary Completion 2013-12 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Depression | 1 month after surgery
  The Hamilton Depression Rating Scale (HDRS) scores
General health status | 1 month after surgery
  36-Item Short-From Health Survey (SF-36) scores

SECONDARY OUTCOMES:
MACE | 6 month
  Composite of major adverse cardiac events (MACE) including death, myocardial infarction and/or revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Zhe Zheng, M.D., Ph.D., Principal Investigator — China National Center for Cardiovascular Diseases
Locations (1):
- China National Center for Cardiovascular Diseases, Beijing, Beijing Municipality, China